CLINICAL TRIAL: NCT05441748
Title: The Microbial and Metabolic Impact of Walnut Consumption in Adults With Obesity
Brief Title: Walnut Consumption and Gut Microbiota
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Hannah Holscher, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20164
Record Dates: First submitted 2021-05-06; First posted 2022-07-01 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Obesity; Inflammation
Keywords: Walnuts; gastrointestinal microbiota; bile acid profiles; inflammation; glycemia; insulinemia
MeSH Terms: conditions — Obesity; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention treatment (Experimental): Intervention treatment will contain walnuts and be consumed everyday for 3 weeks.
  Interventions: Other: Walnuts
- Intervention treatment oil (Experimental): Intervention treatment will contain walnut oil in foods and be consumed everyday for 3 weeks.
  Interventions: Other: Walnut Oil
- Control treatment (Placebo Comparator): Intervention treatment will contain corn oil in foods and be consumed everyday for 3 weeks.
  Interventions: Other: Control

INTERVENTIONS:
Other: Walnuts — The intervention treatment will contain walnuts.
  Arms: Intervention treatment
Other: Walnut Oil — The intervention treatment will contain walnut oil.
  Arms: Intervention treatment oil
Other: Control — The control treatment will contain corn oil.
  Arms: Control treatment

SUMMARY:
Obesity is a growing health issue that effects the majority of adults in the United States. Prevalence of other metabolic diseases are increased in obese adults, including systemic inflammation. There is emerging evidence that the gut microbiota have a mediating role in controlling inflammation by producing butyrate when ingested fiber is fermented. Since these microbes are modifiable by diet, the investigators plan to introduce walnuts to the diets of participants with obesity because they are rich in fiber and unsaturated fatty acids. The purpose of this study is to understand the impacts of walnut consumption on the gut microbiota and the effect they have on bile acid profiles and systemic inflammation. The investigators intention is to identify how these walnut-derived molecules influence Faecalibacterium spp., a butyrate producing microbe. Increased levels of butyrate have shown to decrease secondary bile acids and decrease inflammation.

ELIGIBILITY:
Inclusion Criteria:

Participants will include adults ages 25-75 years BMI of > 30 kg/m2 Ability to drop-off fecal sample within 15 minutes of defecation

Exclusion Criteria:

* Walnut allergy or intolerance
* Food allergies or intolerances
* Prior diagnosis of metabolic or gastrointestinal disease (cardiovascular disease and type 1 or type 2 diabetes, chronic constipation, diarrhea, Crohn's disease, celiac disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers, hepatitis, HIV, cancer, etc.)
* Women that are pregnant, had a baby within the last 12 months, or lactating
* Individuals that smoke, use tobacco, abuse drugs, or consume > 2 alcoholic beverages per day.
* > 5% weight change in the past month or > 10% change in the past year
* Oral antibiotics during the previous 6 weeks
* Fasting blood glucose >126 mg/dL, blood pressure >160/100 mm Hg, elevation in serum transaminases (i.e. >3 times the upper limit of normal) or with evidence of liver disease, including primary biliary cirrhosis or gallbladder disease, constipation, are currently taking lipid-lowering medications, oral hypoglycemic agents, or insulin, or certain medications (laxatives, bile acid sequestrants, and opiates)
* History of malabsorptive or restrictive bariatric surgeries (e.g., gastric bypass, sleeve gastrectomy, adjustable gastric band) or gall bladder removal surgery.
* Are unable to consume the experimental meals/snacks.
* Participants who have donated blood within the last 8 weeks
* Recent diagnosis of anemia
* Concurrent enrollment in another dietary, exercise, or medication study

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Fecal Microbial Species | Fecal samples will be collected at the end of each 3 week condition.
  Abundances of fecal Faecalibacterium spp. and Roseburia spp measured using metagenomic sequencing in walnut and walnut oil vs. control.
Concentration of fecal bile acids | Fecal samples will be collected at the end of each 3 week condition.
  Fecal bile acid concentrations measured using HPLC in walnut and walnut oil vs. control

SECONDARY OUTCOMES:
Fecal Microbial Metabolites | Fecal samples will be collected once at the end of each 3 week condition.
  Concentrations of fecal microbial metabolite (phenol/indoles, short chain fatty acids, and ammonia) concentrations measured using GC-MS in walnut and walnut oil in comparison to a control (corn oil)

OTHER OUTCOMES:
Fecal Microbiome | Fecal samples will be collected at the end of each 3 week condition.
  Relative abundance of microbial genes and genera measured using metagenomic sequencing of extracted fecal DNA to compare abundances between walnut, walnut oil, and corn oil.
Inflammatory markers | Blood samples will be collected at the end of each 3 week condition.
  LPS-binding protein and inflammatory markers (CRP and TNFa) concentrations in walnut and walnut oil vs. control (corn oil)
Serum bile acid profiles | Blood samples will be collected during a mixed-meal tolerance test that occurs at the end of each 3 week condition.
  Serum bile acid concentrations will be measured using LC-ESI-MS/MS to compare concentrations between walnut and walnut oil and control (corn oil)
Mixed-meal tolerance test | At the end of each 3 week condition.
  Blood glucose and insulin concentrations and area under the curve will be measured in blood during a mixed meal tolerance test that includes a standard glucose beverage and the respective walnut, walnut oil, or corn oil treatment.
Intestinal permeability | 24-hour urine collections will occur at the end of each 3 week condition
  Intestinal permeability will be measured using a orally ingested sugar substitutes. 24-hour urinary appearance of the sugars will be quantified using GC-MS.

CONTACTS AND LOCATIONS:
Locations (1):
- Hannah Holscher, Urbana, Illinois, United States